CLINICAL TRIAL: NCT00837291
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of the Efficacy and Safety of Daily CF101 Administered Orally for 12 Weeks to Patients With Osteoarthritis of the Knee
Brief Title: A Study of the Efficacy and Safety of CF101 to Patients With Osteoarthritis of the Knee
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The company has decided not to conduct the study
Sponsor: Can-Fite BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF101-221OA
Record Dates: First submitted 2009-02-03; First posted 2009-02-05 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis; knee; CF101
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — CF101; N(6)-(3-iodobenzyl)-5'-N-methylcarboxamidoadenosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CF101 1 mg BID (Experimental)
  Interventions: Drug: CF101
- Placebo (Placebo Comparator): Placebo tablets BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CF101 — CF101 tablets 1 mg BID
  Other Names: IB-MECA
  Arms: CF101 1 mg BID
Drug: Placebo — Placebo tablets BID
  Other Names: Inactive tablets
  Arms: Placebo

SUMMARY:
This study will test the effectiveness of CF101 in treating the symptoms of osteoarthritis (OA) of the knee. Eligible patients will be given either CF101 or matching placebo tablets and their symptoms will be evaluated over the 12 week treatment period.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, placebo-controlled, parallel-group study in which patients with knee OA will be randomized to either CF101 1 mg or matching placebo tablets every 12 hours and followed for 12 weeks on treatment. For patients with bilateral knee involvement, only 1 knee will be selected for evaluation, namely, the most severely involved knee that meets study criteria (the "index knee"). Screening examinations will occur within 1 month prior to dosing. Washout of non-specific non-steroidal anti-inflammatory drugs (nsNSAIDs) and cyclo-oxygenase-2 (COX-2) inhibitors will occur prior to dosing, and must be followed by requalification before dosing. Disease activity will be assessed using changes from baseline in Patient's Global Assessment (PGA) and Investigator's Global Assessment (IGA) scores, and the Western Ontario and McMaster Universities Osteoarthritis (WOMAC) index and subscales for pain, physical function, stiffness, according to the Outcome Measures in Rheumatology Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) criteria. Assessments will take place at Screening, Baseline (Week 0), and at Weeks 2, 4, 8, 12, and 14.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 40 years or above
* Clinical evidence of knee OA, as indicated by:

  * Pain requiring treatment with NSAID or coxib medication for analgesia for at least 6 months prior to the screening visit, and
  * Pain requiring treatment with NSAID or coxib medication for analgesia on the majority of days during the preceding month
* Radiographic evidence of knee OA, as indicated by findings of Kellgren-Lawrence Grade 2 or 3 within 1 year prior to the screening visit2
* American College of Rheumatology functional class I, II, or III3
* WOMAC pain subscale score ≥40 mm at baseline
* WOMAC function subscale score >20 mm at baseline
* PGA >10 mm at baseline
* In the Investigator's opinion, the ability to understand the nature of the study and any hazards of participation, and to communicate satisfactorily with the Investigator and to participate in, and to comply with, the requirements of the entire protocol
* Negative screening serum pregnancy test for female patients of childbearing potential
* Females of childbearing potential must utilize, throughout the course of the trial, 2 methods of contraception deemed adequate by the Investigator (for example, oral contraceptive pills plus a barrier method)
* All aspects of the protocol explained and written informed consent obtained

Exclusion Criteria:

* Predominant patellofemoral disease
* Concomitant local or systemic inflammatory arthropathy which could confound evaluation of the knee
* Ipsilateral hip or extremity disease which could confound evaluation of the knee
* History of clinical significant trauma or surgery to the index knee
* Arthroscopy to the index knee within 6 months prior to the screening visit
* Corticosteroid, hyaluronic acid, or other intraatricular injection to the index knee within 3 months prior to the screening visit
* Use of chondroitin sulfate and/or glucosamine, or diacerin, within 2 weeks prior to the screening visit
* Concomitant requirement for NSAID, coxib medication, or opioid analgesics (acetaminophen is allowed)
* Use of systemic corticosteroids >10 mg/d of prednisone, or equivalent
* Presence or history of uncontrolled arterial hypertension or symptomatic hypotension
* Significant cardiac arrhythmia or conduction block, congestive heart failure, or any other evidence of clinically significant heart disease; other clinically significant findings on screening electrocardiogram (ECG)
* Hemoglobin level <10.0 gm/dL at the screening visit
* White blood cell count <3000/mm3 at the screening visit
* Platelet count <125,000/mm3 at the screening visit
* Serum creatinine level outside the central laboratory's normal limits at the screening visit
* Liver aminotransferase (ALT and/or AST) levels greater than the upper limit of normal at the screening visit
* Known or suspected immunodeficiency or human immunodeficiency virus positivity
* Pregnancy, lactation, or inadequate contraception as judged by the Investigator
* Participation in another investigational drug or vaccine trial concurrently or within 30 days prior to screening
* History of drug or alcohol dependence
* History of malignancy within the past 5 years (excluding excised basal or squamous cell carcinoma of the skin)
* Diagnosis of Parkinson's Disease
* Significant acute or chronic medical or psychiatric illness that, in the judgment of the Investigator, could compromise patient safety, limit the patient's ability to complete the study, and/or compromise the objectives of the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of responders by OMERACT-OARSI definition | 12 weeks

SECONDARY OUTCOMES:
Safety, as assessed through vital signs, physical examinations, adverse event reporting, clinical laboratory testing, and ECGs | 14 weeks
Change from baseline in total WOMAC score, and pain, physical function, and stiffness subscale scores | 12 weeks
Change from baseline in physician's and patient's global assessments | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Silverman, MD, Study Director — Can-Fite BioPharma Ltd
Locations (1):
- Barzilai Medical Center, Ashkelon, Israel

REFERENCES:
- [Background] Baharav E, Bar-Yehuda S, Madi L, Silberman D, Rath-Wolfson L, Halpren M, Ochaion A, Weinberger A, Fishman P. Antiinflammatory effect of A3 adenosine receptor agonists in murine autoimmune arthritis models. J Rheumatol. 2005 Mar;32(3):469-76. PMID 15742438
- [Background] Bar-Yehuda S, Silverman MH, Kerns WD, Ochaion A, Cohen S, Fishman P. The anti-inflammatory effect of A3 adenosine receptor agonists: a novel targeted therapy for rheumatoid arthritis. Expert Opin Investig Drugs. 2007 Oct;16(10):1601-13. doi: 10.1517/13543784.16.10.1601. PMID 17922624
- [Background] van Troostenburg AR, Clark EV, Carey WD, Warrington SJ, Kerns WD, Cohn I, Silverman MH, Bar-Yehuda S, Fong KL, Fishman P. Tolerability, pharmacokinetics and concentration-dependent hemodynamic effects of oral CF101, an A3 adenosine receptor agonist, in healthy young men. Int J Clin Pharmacol Ther. 2004 Oct;42(10):534-42. doi: 10.5414/cpp42534. PMID 15516022
- See also: Sponsor — http://www.canfite.com
- See also: Additional publications — http://www.canfite.com/publications.html